CLINICAL TRIAL: NCT01999270
Title: Evaluation of FDOPA-PET/MRI in Pediatric Patients With CNS Tumors, A Feasibility Study
Brief Title: Evaluation of FDOPA-PET/MRI in Pediatric Patients With CNS Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201303069
Record Dates: First submitted 2013-11-25; First posted 2013-12-03 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-10

CONDITIONS: Astrocytoma, Oligoastrocytoma, Mixed; Ganglioneuroma; Glioma; Ganglioglioma; Glioblastoma Multiforme Glioma
MeSH Terms: conditions — Astrocytoma; Ganglioneuroma; Glioma; Ganglioglioma | interventions — Irinotecan; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Irinotecan, Bevacizumab and FDOPA-PET/MRI imaging (Experimental): Irinotecan can be removed from the treatment plan at the discretion of the healthcare provider.
  Interventions: Drug: Irinotecan; Drug: Bevacizumab; Device: FDOPA-PET/MRI imaging

INTERVENTIONS:
Drug: Irinotecan — Irinotecan IV over 90 minutes on Days 1, 15, and 29 of each cycle (except Cycle 1, when it will be started on Day 29)
  Note: Irinotecan can be removed from the treatment plan at the discretion of the healthcare provider.
  Other Names: Camptosar®; CPT-11
Drug: Bevacizumab — Bevacizumab will be given intravenously AFTER the irinotecan infusion is complete on Days 1, 15, and 29 of each cycle. The first dose will be given over 90 minutes, but doses after that may be given over 30-60 minutes.
  Other Names: Avastin®
Device: FDOPA-PET/MRI imaging — FDOPA-PET/MRI imaging Baseline (before beginning Cycle 1 treatment) Cycle 1, Day 29 (before receiving your treatment with bevacizumab) and end of treatment or time of relapse

SUMMARY:
To determine if FDOPA-PET/MRI imaging can predict response to treatment of bevacizumab.

DETAILED DESCRIPTION:
Evaluate the feasibility of using FDOPA-PET/MRI pediatric patients with CNS tumors. Positive results in this small study would provide the data needed to expand the study to validate the use in a larger population of pediatric patients. Validating the use of FDOPA-PET imaging as an early predictor for response to anti-angiogenic therapy could greatly impact the standard of care for treating and evaluating pediatric brain tumors and provide a useful biomarker for assessing experimental therapeutics.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have histological verification of one of the eligible diagnosis listed below. Biopsy is required at time of diagnosis, with the exception of optic pathway tumors. Patients with spinal cord disease are eligible if they have a lesion >1 cm in 2 dimensions. The following histologies are eligible:

  * Astrocytoma variants: fibrillary, protoplasmic, mixed
  * Pilocytic astrocytoma, including pilomyxoid variants
  * Pleomorphic xanthoastrocytoma
  * Infantile desmoplastic astrocytoma
  * Ganglioneuroma
  * Oligodendroglial tumor
  * Mixed glioma (including oligoastrocytoma)
  * Anaplastic astrocytoma
  * Anaplastic oligoastrocytoma
  * Anaplastic oligodendroglioma
  * Anaplastic ganglioglioma
  * Glioblastoma multiforme (including giant cell and gliosarcoma types)
  * Medulloblastoma
  * Ependymoma
  * Other rare malignant CNS tumors (i.e., pineal blastoma, small cell astrocytoma, etc.)
* Patient must be ≤ 21 years of age at time of study enrollment.
* Patient must have measurable residual disease, defined as tumor that is measurable in two perpendicular diameters on MRI. Diffuse leptomeningeal disease is not considered measurable.
* Patient must have a Lansky or Karnofsky performance of >40% corresponding to ECOG categories 0, 1, or 2. Karnofsky will be used for patients >16 years of age and Lansky for patients <16 years of age. Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
* Patient must have a life expectancy of >8 weeks.
* Patient must have fully recovered from the acute toxic effects of all prior chemotherapy or radiation prior to entering this study.
* Patient must have recovered from any surgical procedure before enrolling on this study.
* Hypertensive patients are eligible provided the hypertension is well controlled (95th percentile for age and height if patient ≤17 years) on stable doses of medication. (See Appendices I and II for tables of blood pressure based on age and gender).
* Patients receiving corticosteroids are eligible provided the dose is stable or decreasing for at least 7 days.
* Patient must have adequate bone marrow function (including status post-SCT) defined as:

  1. Peripheral absolute neutrophil count (ANC) ≥1000/uL (must not have received G-CSF within the prior 7 days)
  2. Platelet count ≥ 100,000/uL (transfusion independent)
  3. Hemoglobin ≥ 8.0 gm/dL (may receive pRBC transfusions)
* Patient must have adequate renal function defined as:

  1. Creatinine clearance or radioisotope GFR ≥70ml/min/1.73 m2 or
  2. A serum creatinine based on age/gender as follows:

     * 1 month to < 6 months, male max 0.4, female max 0.4
     * 6 months to < 1 year, male max 0.5, female max 0.5
     * 1 to <2 years, male max 0.6, female max 0.6
     * 2 to < 6 years, male max 0.8, female max 0.8
     * 6 to <10 years, male max 1.0, female max 1.0
     * 10 to <13 years, male max 1.2, female max 1.2
     * 13 to <16 years, male max 1.5, female max 1.4

       * 16 years, male max 1.7, female max 1.4
* Urine protein should be screened by dipstick analysis. If protein ≥ 2+ on dipstick, then Urine Protein Creatinine (UPC) ratio should be calculated. If UPC ratio >1, 24-hour urine protein should be obtained and the level should be <1000 mg/24 hours for patient enrollment.

Note: UPC ratio of spot urine is an estimation of the 24 hour urine protein excretion- a UPC ratio of 1 is roughly equivalent to a 24-hour urine protein of 1 gm. UPC ratio is calculated using of the following formulae:

[urine protein]/[urine creatinine] - if both protein and creatinine are reported in mg/dL [(urine protein x 0.088]/[urine creatinine] - if urine creatinine is reported in mmol/L

* Patient must have adequate liver function defined as:

  1. Total bilirubin ≤1.5x upper limit of normal for age (ULN)
  2. SGPT (ALT) ≤ 2.5 x the upper limit of normal (ULN) for age
* Patients with a seizure disorder are eligible if well-controlled on anticonvulsants. If on a non-enzyme inducing anticonvulsant, the irinotecan dose will be adjusted as outline in treatment plan.
* Sexually active patients of childbearing potential must agree to use an effective method of contraception during the study and for at least 6 months after the completion of bevacizumab therapy.
* Patient or legally authorized representative must be able to understand and willing to sign a written informed consent document.

Exclusion Criteria:

* Patient must not have had myelosuppressive chemotherapy ≤ 3 weeks prior to entry onto this study (or 6 weeks if prior nitrosourea).
* Patient must not have had any anti-neoplastic biologic agent ≤7 days prior to entry onto this study (or at least 3 half-lives for biologic agents with a long half-life).
* Patient must not have received craniospinal radiotherapy or involved field radiotherapy to the local tumor (and/or tumor designated as "measurable" for protocol purposes) ≤ 24 weeks prior to study entry; focal radiation to areas of symptomatic metastatic disease must not be given within 14 days of study entry.
* Patient must not have received bevacizumab, or other anti-VEGF inhibitor in the last 3 months.
* Patient must not require a major surgical procedure ≤ 21 days prior to beginning therapy.
* Patient must not require an intermediate surgical procedure ≤14 days prior to beginning therapy.
* Patient must not require a minor surgical procedure (i.e., Broviac line or infusaport placement) ≤ 7 days prior to beginning therapy, and the wound must be healed prior to initiation of therapy.
* There should be no anticipation of need for major surgical procedures during the course of the study.
* Patient must not have received any growth factors ≤7 days of entry onto this study.
* Patient must not be taking NSAIDS, clopidogrel, dipyridamole, or aspirin therapy >81 mg/day.
* Patient must not have a serious or non-healing wound, ulcer, or bone fracture.
* Patient must not require sedation for imaging purposes.
* Patient must not be receiving an investigational drug.
* Patient must not be receiving any other anti-cancer agent.
* Patient must not have an uncontrolled infection.
* Patient must not have a history of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess ≤ 6 months prior to study entry.
* Patient must not have a known bleeding diathesis or coagulopathy.
* Patient must not have had significant vascular disease (e.g., Moya-Moya, aortic aneurysm requiring surgical repair, deep venous or arterial thrombosis) ≤ 6 months prior to study entry.
* Patient must not have a known thrombophilic condition (i.e. protein S, protein C or antithrombin III deficiency, Factor V Leiden, Factor II G20210A mutation, homocysteinemia, or antiphospholipid antibody syndrome). Testing is not required in patients without a thrombophilic history.
* Patient must not have evidence of a new CNS hemorrhage greater than 0.5cm on baseline MRI obtained ≤ 14 days prior to study enrollment.
* Patient must not have a history of stroke, myocardial infarction, transient ischemic attack (TIA), severe or unstable angina, peripheral vascular disease, or grade II or greater congestive heart failure ≤ 6 months prior to study entry.
* Patient must not have serious and inadequately controlled cardiac arrhythmia
* Patient must not be pregnant or breastfeeding.
* Patient must not have a known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies.
* Patient must not be known to be HIV-positive on combination antiretroviral therapy because of the potential for pharmacokinetic interactions with study therapy. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy.
* Patient must not have any contraindications to MRI imaging including implanted medical devices and metal objects which may be adversely affected by MRI imaging. All subjects will be required to complete a standard MRI screening form prior to imaging.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2013-04; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
FDOPA-PET/MRI imaging | 1 year
  The imaging is evaluated: (a) the uptake of PET tracer FDOPA measured by average and maximal standardized uptake values (SUVs) as well as tumor to normal brain ratios; and (b) tumor volumes defined by MRI signal abnormality.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Gauvain, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu